CLINICAL TRIAL: NCT04291014
Title: A Dose Selection Trial of Light Therapy for Impaired Sleep in Parkinson's Disease
Brief Title: Light Therapy for PD - Dose Selection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aleksandar Videnovic, MD, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NN110 1U01NS114001
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease; Sleep Disorder; Fatigue
Keywords: Parkinson Disease; Light therapy
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: This is a 16-week, randomized, phase II, parallel-group, dose-selection clinical trial of LT in participants with PD and co-existing sleep disruption using a comparative selection trial design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BWLT once daily (Experimental): Participants in this arm will receive bright white light therapy daily once a day (in the evening)
  Interventions: Device: SunRay Light Boxes
- BWLT twice daily (Experimental): Participants in this arm will receive bright white light therapy daily twice a day (morning and evening).
  Interventions: Device: SunRay Light Boxes
- BWLT weekly (Experimental): Participants in this arm will receive bright white light therapy once weekly (in the evening).
  Interventions: Device: SunRay Light Boxes
- DRLT twice daily (Experimental): Participants in this arm will receive dim red light twice daily (morning and evening).
  Interventions: Device: SunRay Light Boxes

INTERVENTIONS:
Device: SunRay Light Boxes — SunRay light boxes will be used to administer the light therapy.

SUMMARY:
This study aims to determine the most effective dose of light therapy to improve sleep in people with Parkinson's Disease. Four groups of participants will receive bright-white or dim-red light therapy at different times throughout the day.

DETAILED DESCRIPTION:
This is a 16-week, randomized, phase II, parallel-group, dose-selection clinical trial of LT in participants with PD and co-existing sleep disruption using a comparative selection trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD as defined by the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease;
2. PD Hoehn and Yahr stage 2-4;
3. A score of 2 (mild) or above on the Sleep Problems question of the MDS-UPDRS Part 1;
4. Stable dose of all PD medications for at least 30 days prior to randomization;
5. Willingness to wear an Actiwatch and complete daily sleep logs;
6. Age 45 or above

Exclusion Criteria:

1. Atypical or secondary forms of parkinsonism;
2. Co-existent significant sleep apnea at screening, as determined by the PI's clinical assessment; adequately treated sleep apnea, as assessed by sleep apnea machine download (CPAP download) will be permitted;
3. Co-existent symptomatic restless legs syndrome (RLS) (as assessed by the International Classification of Sleep Disorders (ICDS) diagnostic criteria for RLS) at screening;
4. Cognitive impairment as determined by a Mini Mental State Examination score <25 at screening;
5. Presence of moderate depression defined as a Beck Depression Inventory II (BDI-II) score ≥20 at screening;
6. Current untreated hallucinations or psychosis (drug-induced or spontaneous) with a score of 2 or above on the Hallucinations and Psychosis question of the MDS-UPDRS Part 2;
7. Use of hypno-sedative drugs for sleep or stimulants, unless the participant has been on a stable dose for at least 60 days prior to the screening;
8. Ongoing or recent (within 30 days prior to screening) Cognitive Behavioral Therapy for Insomnia;
9. Use of antidepressants, unless the participant has been on a stable dose for at least 60 days prior to the screening;
10. Work hours between 10 PM and 6 AM, within 60 days prior to randomization or anticipated during the 16 weeks after screening;
11. Travel between 3 or more time zones within 45 days prior to study screening or anticipated such travel during the 16 weeks after screening;
12. Unstable or serious medical illness;
13. History of significant eye trauma or disease, retinopathy, or cataract Grade 4 that would significantly affect transmission or processing of light through either eye;
14. Current use, use at any time during study participation, or use within the 30 days prior to screening of photosensitizing or other medications that in the opinion of the investigator would interfere with the safety of the participant during the trial, including: amiodarone, porfimer, psoralens, chlorpromazine, quinidine, demeclocycline, temoporfin, tetracycline, fleroxacin, oral isoretinoin, voriconazole, nalidixic acid, thioridazine, St. John's wort, ofloxacin, and piroxicam;
15. Pregnant women will be excluded from participation; if a participant is pre-menopausal, a urine pregnancy test will be conducted at randomization to determine eligibility.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
PDSS-2 | 8 weeks
  The PDSS-2 is a 15-question instrument designed to simultaneously capture the multidimensional aspects of sleep-related problems and changes in sleep quality.

SECONDARY OUTCOMES:
PFS-16 | 8 weeks
  The PFS-16 is a patient-rated scale that measures fatigue. The scale allows the measurements of the presence of fatigue (seven items) and its impact on daily function (nine items).

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of Alabama, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC Irvine, Irvine, California
  - UC Davis, Sacramento, California
  - Yale University, Fairfield, Connecticut
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Weill Cornell, New York, New York
  - Mount Sinai - Icahn School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stonybrook, Stony Brook, New York
  - SUNY Upstate, Syracuse, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
This trial will follow the NINDS policy for data sharing.

REFERENCES:
- [Background] Willis GL, Turner EJ. Primary and secondary features of Parkinson's disease improve with strategic exposure to bright light: a case series study. Chronobiol Int. 2007;24(3):521-37. doi: 10.1080/07420520701420717. PMID 17612949
- [Background] Paus S, Schmitz-Hubsch T, Wullner U, Vogel A, Klockgether T, Abele M. Bright light therapy in Parkinson's disease: a pilot study. Mov Disord. 2007 Jul 30;22(10):1495-1498. doi: 10.1002/mds.21542. PMID 17516492
- [Background] Terman M, Terman JS. Bright light therapy: side effects and benefits across the symptom spectrum. J Clin Psychiatry. 1999 Nov;60(11):799-808; quiz 809. PMID 10584776
- [Background] Gallin PF, Terman M, Reme CE, Rafferty B, Terman JS, Burde RM. Ophthalmologic examination of patients with seasonal affective disorder, before and after bright light therapy. Am J Ophthalmol. 1995 Feb;119(2):202-10. doi: 10.1016/s0002-9394(14)73874-7. PMID 7832227
- [Background] Videnovic A, Klerman EB, Wang W, Marconi A, Kuhta T, Zee PC. Timed Light Therapy for Sleep and Daytime Sleepiness Associated With Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2017 Apr 1;74(4):411-418. doi: 10.1001/jamaneurol.2016.5192. PMID 28241159
- [Background] Trenkwalder C, Kohnen R, Hogl B, Metta V, Sixel-Doring F, Frauscher B, Hulsmann J, Martinez-Martin P, Chaudhuri KR. Parkinson's disease sleep scale--validation of the revised version PDSS-2. Mov Disord. 2011 Mar;26(4):644-52. doi: 10.1002/mds.23476. Epub 2011 Feb 10. PMID 21312275
- [Background] Brown RG, Dittner A, Findley L, Wessely SC. The Parkinson fatigue scale. Parkinsonism Relat Disord. 2005 Jan;11(1):49-55. doi: 10.1016/j.parkreldis.2004.07.007. PMID 15619463